CLINICAL TRIAL: NCT05546047
Title: A Multicenter, Comparative Safety and Efficacy Study of ACTHar Gel Alone or in Combination With Oral Tacrolimus to Reduce Urinary Proteinuria in Patients With Idiopathic DNAJB9 Positive Fibrillary Glomerulopathy
Brief Title: A Study of Acthar Gel Alone or With Tacrolimus to Reduce Proteinuria in Fibrillary Glomerulopathy Patients
Acronym: FACT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: NephroNet, Inc. (Other)
Collaborators: Mallinckrodt (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN-002
Record Dates: First submitted 2022-08-23; First posted 2022-09-19 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Fibrillary Glomerulonephritis
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Intervention Model Description: A 12-month treatment with combination Acthar gel and Tacrolimus therapy will be superior to Acthar gel therapy alone in lowering urinary protein to creatinine ratios in patients with Fibrillary glomerulonephritis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment with Acthar gel (Active Comparator): Group 1 - (17 patients) Acthar gel 80 units 2 times a week alone for 12 months of therapy.
  Interventions: Drug: Acthar Gel 80 UNT/ML Injectable Solution
- Treatment with combination Acthar gel and Tacrolimus therapy (Active Comparator): Group 2 - (17 patients) Acthar get 80 units 2 times a week plus oral Tacrolimus 1.0 mg two times a day titrated to trough Tacrolimus levels between 4-6 ng/ml
  Interventions: Drug: Acthar Gel 80 UNT/ML Injectable Solution

INTERVENTIONS:
Drug: Acthar Gel 80 UNT/ML Injectable Solution — Follow up and observation for 12 months off Acthar gel or Acthar gel and Tacrolimus
  Other Names: Tacrolimus 1.0 mg

SUMMARY:
A Multicenter, Comparative Safety and Efficacy Study of Acthar gel alone or in combination with oral Tacrolimus to reduce urinary proteinuria in patients with idiopathic DNAJB9 Positive Fibrillary glomerulopathy.

DETAILED DESCRIPTION:
A Multicenter, Comparative Safety and Efficacy Study of Acthar gel alone or in combination with oral Tacrolimus to reduce urinary proteinuria in patients with idiopathic DNAJB9 Positive Fibrillary glomerulopathy. This study will be a multi-center, prospective, randomized, open-labeled intervention trial of 34 patients randomized to 52 weeks of ACTHar gel alone or Acthar gel plus oral Tacrolimus.

ELIGIBILITY:
Inclusion Criteria:

* Male/Female age > 18
* Biopsy proven Fibrillary glomerulonephritis within 3 years of study randomization
* Stable Maximum Renin-Angiotensin-Aldosterone System inhibition times 4 weeks prior to randomization Note: Maximum RAAS inhibition will be left to the discretion of the site Principal Investigator
* Estimated Glomerular Filtration Rate > 25 mls/min calculate by the Chronic Kidney Disease-EPI formula
* Protein/creatinine ratio > 2000 mg/gm 5) Note: If protein/creatinine less than 2000 mg/gm, a formal 24- hour urine collection for total protein can be performed. The total 24-hour protein will need to >/= 2000mg.
* Blood pressure targeted to < 140/90 at the time of randomization
* Patients with Monoclonal Gammopathy without history of myeloma will be eligible.
* Patients with monoclonal staining for fibrillary fibers will be excluded
* Patients with Type II non-insulin dependent diabetes will be eligible provided the renal biopsy does not show nodular Kimmelstiel Wilson lesions

Exclusion Criteria:

* Patients with MGUS and history of myeloma will not be eligible
* Patients with active viral production of either hepatitis B or C as evidence by historical polymerase chain reaction test positive for active viral shedding
* HIV seropositivity
* Renal biopsy data with > 50% Interstitial Fibrosis
* Patient with active or a known history lymphoma
* Patients with insulin dependent diabetes mellitus will be excluded Note: patients with Type II diabetes mellitus that are well controlled without the need for insulin will be eligible for the study.
* Patients with Type II non-insulin dependent diabetes will be eligible provided the renal biopsy does not show nodular Kimmelstiel Wilson lesions.
* Patients receiving steroids, mycophenolate mofetil, cyclophosphamide, Azathioprine or other immunosuppressive agent with 4 weeks of study randomization Note: Washout of these medications will be allowed at the screening visit
* Patients having received Rituximab or B cell modifying biologic therapy within 6 months of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2019-03-14 (Actual); Primary Completion 2023-10-27 (Estimated); Study Completion 2024-10-27 (Estimated)

PRIMARY OUTCOMES:
The change in UP/CR ratio with treatment of Acthar gel 80 units subcutaneous 2 times a week alone | 12 months
  The change in protein/creatinine ratio in patients with biopsy proven Fibrillary after 12 months of treatment with treated with Acthar gel (80 units subcutaneous 2 times a week) alone
The change in UP/CR ratio with treatment of Acthar gel 80 units subcutaneous 2 times a week in combination with oral Tacrolimus | 12 months
  The change in protein/creatinine ratio in patients with biopsy proven Fibrillary after 12 months of treatment with treated with Acthar gel 80 units 2 times a week subcutaneous week in combination with oral Tacrolimus 1.0 mg orally two times a day.

SECONDARY OUTCOMES:
The relative change in protein/creatinine ratio at 24 months | 24 months
  The relative change in protein/creatinine at 24 months (12 months after stopping both Acthar and Tacrolimus) in the Acthar gel group and the Acthar gel plus Tacrolimus group.
Percentage of patients complete or partial response | 12 months
  The percentage of patients in the Acthar gel alone versus Acthar gel + Tacrolimus group that achieves complete, partial or clinical responses after 12 months of therapy
The change in Estimated Glomerular Filtration Rate | 24 months
  The change in Estimated Glomerular Filtration Rate between the Acthar gel and Acthar Gel plus Tacrolimus groups after 24 months of treatment with Acthar gel alone or in combination with oral Tacrolimus. In addition, we will also compare the relative change in eGFR between those patients receiving Acthar gel alone with those randomized to combination therapy.
To compare the change in urinary biomarkers of Urinary VEGF 121, 165 189, and206, Urinary MCP-1, Urinary Synaptopodin, Urinary TGF-beta, Urinary Podocalyxin, and Urinary Nephrin | 12 months
  To compare the change in urinary biomarkers at baseline and after 12 months of treatment with Acthar gel alone or in combination with Tacrolimus. The patients urinary biomarker levels after 12 months of therapy will be compared between the Acthar gel alone group and Acthar gel plus Tacrolimus group.
  1. Urinary VEGF 121, 165 189, and206
  2. Urinary MCP-1
  3. Urinary Synaptopodin
  4. Urinary TGF-beta
  5. Urinary Podocalyxin
  6. Urinary Nephrin

OTHER OUTCOMES:
To determine if patients with concurrent Type II diabetes mellitus resulted in hyperglycemia, increased proteinuria, loss of renal function or led to immunosuppressive therapies | 24 months
  To determine whether Acthar gel therapy resulted in hyperglycemia in patients with concurrent Diabetes and whether that led to early termination from the study. We will also determine whether the presence of diabetes led to increased proteinuria over time, led to more rapid decline in renal function and altered the response to immunosuppressive therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Whitson, BS, Study Director — NephroNet, Inc.; James Tumlin, MD, Principal Investigator — NephroNet, Inc.
Locations (5):
- United States (5):
  - Stanford University, Stanford, California
  - University of Colorado Anschutz Medical Department of Medicine Division of Renal Diseases and Hypertension, Aurora, Colorado
  - Georgia Nephrology DBA Georgia Nephrology Research Institute, Lawrenceville, Georgia
  - Columbia University Research Dept of Nephrology, New York, New York
  - Northeast Clinical Research Center, Bethlehem, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2019-03-14): https://cdn.clinicaltrials.gov/large-docs/47/NCT05546047/Prot_000.pdf